CLINICAL TRIAL: NCT04077138
Title: Transgender Youth and PrEP: PK, Safety, Uptake & Adherence
Brief Title: Transgender Youth and PrEP: PK, Safety, Uptake & Adherence - Intervention Development
Status: Completed | Type: Observational
Sponsor: Hektoen Institute for Medical Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01MH114753-2; R01MH114753 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2019-09-04 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS; Gender; Behavior and Behavior Mechanisms
Keywords: Transgender; Pre-exposure Prophylaxis (PrEP); HIV Prevention; Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC); Cross-sex Hormone Therapy; Adherence; Behavior Change; Gender Affirmation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Focus Groups: Ten focus groups with transgender women and transgender men will be conducted. . The structure of the focus groups will utilize an interactive "Rapid Approach", which differs from traditional focus groups by asking fewer questions and tightly focusing on specific areas of inquiry.
- In-Depth Interviews: Participants for the IDIs, 10-15 TW and TM, will be selected from among Phase 1 participants. We will create a purposive sample that represents a range of experiences that occurred during Phase 1.

SUMMARY:
To address the critical scientific gaps in PrEP safety for transgender youth and to plan for appropriate implementation of PrEP in transgender youth communities, the study will be conducted in 3 integrated phases. In Phase 1, a pharmacokinetic (PK) study exploring the interactions of cs-HT for both TW and TM youth on TDF/FTC will be conducted. Simultaneously, in Phase 2, ethnographic data via focus groups (FGs) and in-depth interviews (IDIs) to inform the development of a tailored intervention to improve uptake and adherence to PrEP for transgender youth will be collected. In Phase 3, a small demonstration trial of PrEP use in transgender youth, utilizing the ethnographically developed intervention to improve uptake and adherence, while also monitoring renal and bone safety outcomes will be implemented.

The project has the following important specific aims:

Aim 1: To evaluate the differential PK of TDF/FTC in a cohort of transgender youth on cs-HT by conducting a PK trial of daily TDF/FTC among 24 TW taking estradiol and 24 TM taking testosterone (ages 15-24 years) using video-based directly observed therapy (DOT) to insure daily adherence and maximize drug exposure.

Aim 2: To develop a culturally, developmentally, and gender-affirmative intervention to increase uptake of and adherence to PrEP among TW and TM youth that is grounded in theory (Information-Motivation-Behavioral Skills Model of Behavior Change, Gender Affirmation, Empowerment Theory) and incorporates the PK data from Aim 1. Investigators will conduct FGs with young TW (N=20-30) and TM (N=20-30) and conduct IDIs with participants from the PK study (Total N=10-14). Investigators will solicit continuous input and feedback from TW and TM on the project's Youth Advisory Board.

Aim 3: To conduct a small randomized controlled trial within a PrEP demonstration project comparing the newly developed intervention with standard of care (SOC) in TW (N=50) and TM (N=50) ages 15-24 years.

DETAILED DESCRIPTION:
Transgender women (TW) are one of the most vulnerable populations for acquiring HIV infection, and the scant available data on transgender men (TM) suggests they are also at risk. TW have accounted for only 0.2% of all participants in bio-behavioral HIV prevention trials using pre-exposure prophylaxis (PrEP), and TM have typically not been included. TW and TM adolescents have received even less attention in PrEP trials.

Although tenofovir disoproxil fumarate/emtricitabine (TDF/FTC), the FDA-approved PrEP drug, would not be expected to interact with cross-sex hormone therapy (cs-HT; estradiol and testosterone) based on known mechanisms and data from studies with hormonal contraceptives, there are no data that prove this. Given this lack of data, TW and TM youth on cs-HT have decreased PrEP uptake and adherence due to concerns that PrEP may reduce the effectiveness of cs-HT. To address these critical scientific gaps in PrEP safety for transgender youth and to plan for appropriate implementation the investigators propose the following study in 3 integrated phases. In Phase 1, investigators will conduct a PK study exploring the interactions of cs-HT for both TW and TM on TDF/FTC. Simultaneously, in Phase 2, investigators will collect ethnographic data via focus groups and in-depth interviews to inform the development of a tailored gender-affirmative intervention to improve uptake and adherence to PrEP in transgender youth. In Phase 3, investigators will conduct a small demonstration trial of PrEP use in TW and TM youth, utilizing the ethnographically developed intervention to improve uptake and adherence, while also monitoring renal and bone safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Able to provide informed consent in English
* Self-reports HIV transmission risk behavior including one or more of the following: a) condomless anal or vaginal intercourse, b) 3 or more sexual partners in the past 3 months, c) any diagnosis by self-report of a STI in the past 12 months, and e) any history of transactional sex work

Exclusion Criteria:

* Hospitalization within 30 days of study entry (elective procedures okay with team approval)
* Condition (medical, psychological, or social) that, in the opinion of the study investigators, would preclude the participant from completing study-required procedures
* Previous participation in an HIV vaccine study, unless the participant can document placebo arm assignment
* Use of TDF/FTC in the past 3 months

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identification as a transgender individual
Study Population: Transgender women youth and transgender men youth at high-risk of acquiring HIV
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Qualitative Interviews | Year 2
  Focus groups and in-depth interviews with young transgender women and transgender men will combine with PK data from phase 1 to inform the development of a culturally, developmentally, and gender-affirmative intervention to increase uptake of and adherence to PrEP among TW and TM youth.

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Principal Investigator — Cook County Health
Locations (3):
- United States (3):
  - University of Colorado, Denver, Denver, Colorado
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No